CLINICAL TRIAL: NCT07068867
Title: A Protocolled Implementation of Upfront Ultrasound (Sequential Pre-operative Imaging) in Primary Hyperparathyroidism in the Region of Southern Denmark
Brief Title: Upfront Ultrasound for Preoperative Localization in Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Acadre project ID: 23/36379; A5992 (Other Grant/Funding Number: OUH Fund for Pre-graduate Stipends)
Record Dates: First submitted 2025-03-13; First posted 2025-07-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Primary Hyperparathyroidism
Keywords: Parathyroid Diseases; Ultrasound; Preoperative Procedures; Preoperative Localization; Endocrine System Diseases; Hyperparathyroidism; Hyperparathyroidism, Primary
MeSH Terms: conditions — Hyperparathyroidism, Primary; Parathyroid Diseases; Endocrine System Diseases; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary hyperparathyroidism is caused by overactive parathyroid glands, leading to elevated calcium levels in the blood. The standard preoperative imaging includes both a radiation-based imaging modality and conventional ultrasound. However, ultrasound alone is a faster, safer, and more patient-friendly alternative. This study evaluates an upfront ultrasound approach, where patients undergo ultrasound first, and only those with certain findings proceed directly to surgery without additional imaging. Patients with uncertain findings proceed to additional imaging. The study is designed as a prospective cohort with a non-inferiority analysis, aiming to confirm whether upfront ultrasound can achieve an acceptable diagnostic sensitivity. If successful, this approach could reduce patient burden, minimize radiation exposure, and optimize healthcare resources

DETAILED DESCRIPTION:
This study evaluates the implementation of a stepwise approach using upfront ultrasound for localizing pathological parathyroid glands in patients with primary hyperparathyroidism (PHPT).

PHPT is caused by overactive parathyroid glands, leading to excessive amounts of calcium in the blood, which can result in complications such as kidney stones, osteoporosis, cardiovascular disease, and neurological symptoms. The standard preoperative imaging process currently includes both nuclear medicine scans and ultrasound. However, nuclear imaging is time-consuming, exposes patients to radiation, and may not always provide definitive results.

The proposed approach prioritizes ultrasound as the initial localization tool, with additional imaging reserved for cases where ultrasound findings are inconclusive. This method has the potential to reduce unnecessary hospital visits, minimize radiation exposure, and streamline the diagnostic process. The study aims to ensure that this approach maintains high sensitivity for the localization of pathological parathyroid glands, with a target sensitivity of at least 89.5% for correctly identifying diseased parathyroid glands.

Designed as a prospective cohort study, the project will assess patients using ultrasound first, assigning confidence scores (0-3) to determine whether further imaging is necessary. A confidence-score of 3 indicates a high diagnostic confidence. To gain a score of 3, the potential parathyroid adenoma must meet all predefined criteria, i.e. hypoechogenicity, well-defined margins, location at the anatomically expected position, a polar feeding vessel, and a vascular arc. A diagnostic-score of 2 reflects moderate suspicion, where one or two of these key features are missing. A diagnostic-score of 1 suggests low suspicion, typically characterized by a poorly defined structure with no vascular features. Finally, a diagnostic-score of 0 means that no potential adenoma was detected.

Postoperative findings will confirm the accuracy of the preoperative imaging with the histopathological result of the surgically removed specimen(s) combined with biochemical cure at 6 months as the reference standard.

The study aims to benefit both patients and society as it intends to decrease patient exposure to radiation, reduce costs, and reduce the time patients have to take off from work for the purpose of preoperative imaging. One less hospital visit will also reduce the pollution caused by an extra day of transportation to and from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older with primary hyperparathyroidism referred to the Department of ORL, Head and Neck Surgery at Odense University Hospital for parathyroidectomy.

Exclusion Criteria:

* Other causes of hypercalcemia
* Persistent or recurrent hyperparathyroidism.
* Previous surgery to the thyroid or the parathyroid glands.
* Inability to read/speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older with primary hyperparathyroidism referred to the Department of ORL, Head and Neck Surgery at Odense University Hospital for parathyroidectomy.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the sequential imaging regimen (upfront ultrasound) | No residual disease 6 months after surgery
  The primary outcome measure is the sensitivity of the sequential imaging regimen (upfront ultrasound) for localizing one or more pathological parathyroid glands to the correct quadrant of the neck. The reference standard is histopathology combined with biochemical cure.

SECONDARY OUTCOMES:
Primary outcome re-calculated for a theoretical cut-off at "diagnostic confidence score = 2" | No residual disease 6 months after surgery
  The primary endpoint re-calculated with a theoretical cut-off at "diagnostic confidence score=2" as the criteria that leads to surgery without additional imaging.
Primary outcome re-calculated for a theoretical cut-off at "diagnostic confidence score = 1" | No residual disease 6 months after surgery
  The primary endpoint re-calculated with a theoretical cut-off at "diagnostic confidence score=1" as the criteria that leads to surgery without additional imaging.
Per gland sensitivity, specificity, positive and negative predictive value of the sequential imaging regimen | 6 months after surgery
  Per gland sensitivity, specificity, positive and negative predictive value of the sequential imaging regimen
Patients that didn't need supplementary imaging | 6 months post-surgery
  Fractions of patients that didn't need supplementary imaging.
Surgery duration | Immediately after surgery
  Discrepancy between expected and actual duration of surgery.
Unnecessary supplementary imaging | 6 months post-surgery
  Fraction of unnecessary supplementary imaging
Unnecessarily explored quadrants | 6 months post-surgery
  Number of unnecessarily explored quadrants
Complication rate | From surgery until one year after surgery
  Complication rate in terms of recurrent nerve paralysis, post-operative hemorrhage, or permanent hypoparathyroidism
Cure rate | No residual disease 6 months after surgery
  No hyperparathyroid hypercalcemia
Cost | Through study completion, from baseline to 6 months post-surgery
  Cost of ultrasound, parathyroid scintigraphy and parathyroid choline PET/CT
Confounding | Baseline to 6 months post-surgery
  Is the sensitivity influenced by differences in patient age, sex, BMI, adenoma weight, adenoma depth, adenoma diameter, multiple gland disease, preoperative ionized calcium and preoperative PTH?

CONTACTS AND LOCATIONS:
Overall Officials: Sanne H Michaelsen, MD, Principal Investigator — Odense Universitetshospital; Viveque Egsgaard, MD, PhD, Study Chair — Odense Universitetshospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No